CLINICAL TRIAL: NCT03111862
Title: Observational Study on the Safety of Accelerated Rule-out Protocols in Patients Admitted With Chest Pain to a Crowded CPU
Brief Title: Safety of Accelerated Rule-out Protocols in Patients Admitted With Chest Pain to a Crowded Chest Pain Unit (CPU)
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Moritz Biener, Principal Investigator, University Hospital Heidelberg
Other Study IDs: UHHD-BM-004
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Acute Coronary Syndrome; NSTEMI - Non-ST Segment Elevation MI
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Clinical Chemistry, in particular High-sensitivity troponin T
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NSTEMI Rule-Out according to hs-TnT — Rule-Out according to the rapid rule-out protocol of the current ESC Guidelines

SUMMARY:
The aim of this observational study registry is to assess the safety of a Non-ST-elevation myocardial infarction (STEMI) rapid rule-out strategy as proposed by European Guidelines in patients presenting with suspected acute coronary syndrome to the emergency department.

DETAILED DESCRIPTION:
Design: mono-center observational study in a University chest pain unit

Duration: 12 months recruitment period starting June 2016 with end of recruitment July 2017. In the first 6 months assessment of situation, January 2017 introduction of fast protocols, i.e. 0/1 h as standard, observation of trend changes, utilization rates, safety from January 1st until July 2017. Another 90 days follow-up after last patient in.

Background: Several rule-out protocols recommended by 2015 European Society of Cardiology (ESC) guidelines, evidence supported by prospectively validated studies. However, no real life experience with ultilization rates and safety.

Particularly overcrowded emergency departments (EDs) or CPUs are likely to benefit most from fast rule-out protocols in order to discharge a substantial proportion of low risk patients.

Study group: consecutive patients presenting to CPU with suspected acute coronary syndrome (ACS) based on chest pain or chest pain equivalent symptoms

Inclusion criteria: eligible to consent, > 18 years

Exclusion criteria: rule-in, observational zone, chronic hemodialysis, no consent, atrial tachyarrhythmias with chest pain or equivalent.

Data collection on: demographics, rule-out diagnostic protocol (instant cardiac troponin+Copeptin, instant at Limit of Detection, 0-1h, 0-3 h, 0-6 hour, other; time of second sample from admission; turnaround time for first and consecutive sample(s); rates of echo, computed tomography (CT) coronary or CT pulmonary artery, CT chest or CT triple rule-out, chest X-ray, stress test performed or recommended within 3 working days; length of stay in ED, length of stay in hospital including initial referral; rates of admission, discharge or referral; rates of in-hospital percutaneous coronary Intervention (PCI) or coronary artery Bypass graft (CABG), coronary angiography findings based on a definition of obstructive coronary artery disease (CAD) ≥ 50% stenosis.

Specific data: Number of patients seeking attendance in CPU per day (crowding index), GRACE score, secondary risk factors present or not (leftventricular ejection fraction (LVEF) < 40%, glomerular filtration rate< 60 ml/min, Diabetes mellitus, previous myocardial infarction (MI), previous CABG, prior PCI, ST segment depression). Rule-out protocols are stratified by hour ± 30 min, i.e. 0-1 h (±30 min), 0-2 h (±30 min), 0-3 h (±30 min) etc.

Clinical work-up results: stress test before discharge positive or negative, transthoracic echocardiography: wall motion abnormalities, LVEF, valvular heart disease, structural heart disease, Endpoint(s): primary safety endpoint defined as survival free of all-cause death, secondary endpoints: survival free of death or MI, survival free of death/MI/re-hospitalisation for ACS, survival free of death/MI/rehospitalisation for non-elective revascularization

Follow-up: 30 days and 3 months follow-up (FU) for all-cause death, MI, re-hospitalisation for ACS, re-hospitalisation for non-elective PCI or CABG Statistical plan: no sample size calculation, Student´s T-test, ANOVA, Kaplan Meier survival, Cox proportional regression analysis

Milestones: Start immediately after contract for a recruitment period 9/16 - 9/17 (12 months) plus 3 months FU after last patient in. Additional 3 months for completion of files and FU data.

ELIGIBILITY:
Inclusion Criteria:

* eligible to consent
* >18 years

Exclusion Criteria:

* NSTEMI rule-in
* hs-TnT in observational zone
* chronic hemodialysis
* no consent
* atrial tachyarrhythmias with chest pain or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting to CPU with suspected ACS based on chest pain or chest pain equivalent symptoms
Sampling Method: Probability Sample
Enrollment: 3567 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
All-cause death | 30 days and 3 months
  Survival free of all-cause death

SECONDARY OUTCOMES:
Acute Myocardial Infarction | 30 days and 3 months
  Non-STEMI and STEMI
Rehospitalization for Acute Coronary Syndrome | 30 days and 3 months
  Acute Coronary Syndrome including unstable angina, non-STEMI and STEMI
Rehospitalization for nonelective percutaneous coronary intervention | 30 days and 3 months
  Unplanned PCI

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Biener, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- Universtity Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reich C, Yildirim M, Salbach C, Biener M, Lopez-Ayala P, Muller C, Frey N, Giannitsis E. Resolving the observe zone: validation of the ESC 0/3-hour and the APACE criteria for NSTEMI triage. Open Heart. 2025 Mar 28;12(1):e003047. doi: 10.1136/openhrt-2024-003047. PMID 40154974
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Aldous SJ, Allen BR, Apple FS, Babel H, Christenson RH, Cullen L, Di Carluccio E, Doudesis D, Ekelund U, Giannitsis E, Greenslade J, Inoue K, Jernberg T, Kavsak P, Keller T, Lee KK, Lindahl B, Lorenz T, Mahler SA, Mills NL, Mokhtari A, Parsonage W, Pickering JW, Pemberton CJ, Reich C, Richards AM, Sandoval Y, Than MP, Toprak B, Troughton RW, Worster A, Zeller T, Ziegler A, Blankenberg S; ARTEMIS study group. Personalized diagnosis in suspected myocardial infarction. Clin Res Cardiol. 2023 Sep;112(9):1288-1301. doi: 10.1007/s00392-023-02206-3. Epub 2023 May 2. PMID 37131096
- [Derived] Stoyanov KM, Biener M, Hund H, Mueller-Hennessen M, Vafaie M, Katus HA, Giannitsis E. Effects of crowding in the emergency department on the diagnosis and management of suspected acute coronary syndrome using rapid algorithms: an observational study. BMJ Open. 2020 Oct 8;10(10):e041757. doi: 10.1136/bmjopen-2020-041757. PMID 33033102
- [Derived] Giannitsis E, Biener M, Hund H, Mueller-Hennessen M, Vafaie M, Gandowitz J, Riedle C, Lohr J, Katus HA, Stoyanov KM. Management and outcomes of patients with unstable angina with undetectable, normal, or intermediate hsTnT levels. Clin Res Cardiol. 2020 Apr;109(4):476-487. doi: 10.1007/s00392-019-01529-4. Epub 2019 Jul 19. PMID 31325044
- [Derived] Stoyanov KM, Hund H, Biener M, Gandowitz J, Riedle C, Lohr J, Mueller-Hennessen M, Vafaie M, Katus HA, Giannitsis E. RAPID-CPU: a prospective study on implementation of the ESC 0/1-hour algorithm and safety of discharge after rule-out of myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2020 Feb;9(1):39-51. doi: 10.1177/2048872619861911. Epub 2019 Jul 12. PMID 31298551